CLINICAL TRIAL: NCT03109639
Title: A Randomized Prospective Comparison of the New EUS Guided Acquire TM Needle Biopsy vs EUS Guided Fine Needle Aspiration for Suspected Solid Gastrointestinal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EUS01042017
Record Dates: First submitted 2017-04-01; First posted 2017-04-12 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumor; Histological Type of Neoplasm
Keywords: EUS; FNA; FNB; Core Histology
MeSH Terms: conditions — Neoplasms by Histologic Type

STUDY DESIGN:
Intervention Model Description: The participants will be randomised to one of the two groups. The first group will undergo tissue acquisition using the conventional EUS needle. After this, the lesion will be punctured again using the experimental Acquire EUS FNB needle to obtain tissue. In the second group, the experimental Acquire EUS FNB needle will be used first followed by the conventional needle to acquire tissue.
Who Masked: Outcomes Assessor
Masking Description: The pathologist will be blinded to the needle used for specimen collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Active Comparator): This group will undergo tissue acquisition using the conventional EUS-FNA needle followed by the experimental Acquire EUS- FNB needle
  Interventions: Device: Conventional EUS FNA needle; Device: Acquire FNB device
- Group B (Active Comparator): This group will undergo tissue acquisition using the experimental Acquire EUS- FNB needle followed by the conventional EUS-FNA needle
  Interventions: Device: Conventional EUS FNA needle; Device: Acquire FNB device

INTERVENTIONS:
Device: Conventional EUS FNA needle — Participants randomised to Group A will undergo tissues acquisition using the Conventional EUS FNA needle and then crossed over to receive the experimental Acquire EUS- FNB device.
Device: Acquire FNB device — Participants randomised to Group B will undergo tissue acquisition using the experimental Acquire EUS FNB device and then crossed over to receive the conventional EUS FNA needle

SUMMARY:
Endoscopic ultrasound guided fine needle aspiration (EUS-FNA) is the technique of choice to evaluate solid gastrointestinal (GI) lesions. The tissue acquired using this technique is essential for diagnosis of diseases like sub-mucosal masses (GIST), lymphoma, autoimmune pancreatitis and pancreatic cancer. Also the availability of adequate tissue will enable performance of molecular profiling and personalized oncologic therapy. The current needle used for tissue acquisition rarely provides tissue blocks needed for histology assessment. Hence, a better needle device with a good safety profile is needed to solve this technical difficulty. The new AcquireTM fine needle biopsy device could over come this difficulty because of its unique designs. The additional cutting edge surface allows better tissue access and provides core tissue (>90%) for histology. The safety profile of this new device is comparable to the conventional FNA needle thereby making it an ideal device for tissue acquisition.

DETAILED DESCRIPTION:
Endoscopic ultrasound has become the preferred method to characterise gastrointestinal (GI) wall and peri-gastrointestinal masses. A major strength is that it can be used to guide fine needle aspiration (EUS-FNA) of any lesion in the wall or within 5cm from the GI tract. However, EUS-FNA has a major drawback- it rarely able to provide tissue blocks. Thus multiple passes, each of them time consuming, are necessary to obtain adequate cellular samples for cytological analysis. A radically new design of FNA needle (AcquireTM) has recently become available. The needle has an additional cutting edge surface, which allows better tissue access and acquires intact large core samples. The flexibility of the needle permits its use in tortuous anatomy, thereby making it an ideal needle for FNA. The new AcquireTM fine needle biopsy device (FNB) provides core tissue (>90%) for histology. This ability of the needle will enable us to obtain core tissue in fewer passes and make a precise diagnosis. However, at present there is no prospective randomized study to validate this finding.

The investigators hypothesize that the unique cutting system of Acquire TM fine needle biopsy (FNB) device will improve the specimen adequacy of solid intestinal and extra-intestinal lesions by providing a good core tissue for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 21 years
2. All patients with solid lesions (pancreas, lymph nodes, metastasis, liver and sub-epithelial lesions) referred for EUS- FNA
3. Solid lesions confirmed by at least a single investigational modality, mainly CT, MRI or endoscopy
4. Able to comply with the study procedure and provide informed consent.

Exclusion Criteria:

1. Presence of active bleeding
2. Presence of coagulopathy as evidenced by INR>1.5 and platelets <50,000
3. Inability to sample because of intervening blood vessels seen during imaging or EUS.
4. Poor patient tolerance to procedure
5. Concurrent intake of anti-coagulants and thienopyridine (e.g clopidogrel) in patients who require anti-platelet therapy.
6. Pregnancy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Tissue adequacy rate will be measured by assessing for the presence of histological core tissue representative of the lesion in the samples obtained using the two needles | 8 months
  The samples will be analyzed by the blinded pathologist for presence of histological core. Based on the presence of histological core, the sample will be graded optimal or suboptimal. Optimal specimens are those in which the procured material enabled satisfactory assessment of histologic architecture. Suboptimal specimens are those in which the quality of the core is inadequate or unsatisfactory for the assessment of histologic architecture

SECONDARY OUTCOMES:
Quantification of the sample obtained using the two EUS needles will be assessed by measuring the DNA and RNA concentration | 8 months
  Both cell block and core biopsies will be deparafinized and extraction with Qiagen RNA/ DNA kit will be performed. Both DNA and RNA will be quantified by Qubit system
Qualification of the sample obtained using the two needles will be performed by spectroscopic analysis.The ratio of absorbance at 260 nm and 280nm; the ratio of absorbance at 260nm and 230nm will be measured | 8 months
  Spectroscopic analysis will be performed to assess the purity samples. The 260/280 and 260/230 ratios will be measured. A lower ratio may indicate the presence of impurities.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No